CLINICAL TRIAL: NCT00746889
Title: Using Ultrasound to Predict Response to Intraarticular Corticosteroids in Knee Osteoarthritis: A Randomized Placebo-Controlled Clinical Trial
Brief Title: Using Ultrasound to Predict Response to Intraarticular Corticosteroids in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Kenneth Kalunian, University of California San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 051420
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2008-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee; corticosteroids; ultrasound
MeSH Terms: conditions — Osteoarthritis | interventions — Triamcinolone Acetonide; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteroid Injection (Active Comparator): 40 mg of intraarticular triamcinolone acetonide
  Interventions: Drug: triamcinolone acetonide
- Placebo Injection (Placebo Comparator): Intraarticular injection of 0.9% saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: triamcinolone acetonide — single intraarticular injection of 40 mg of triamcinolone acetonide
  Arms: Corticosteroid Injection
Drug: saline — Single intraarticular injection of 1 ml of 0.9% saline
  Arms: Placebo Injection

SUMMARY:
A study using characteristics on ultrasound to predict response to intraarticular steroid injections in patients with knee osteoarthritis. The hypothesis is that patients with inflammation on ultrasound will have a better response to corticosteroid injections compared to patients without inflammation.

ELIGIBILITY:
Inclusion Criteria:

* knee pain
* diagnosis of osteoarthritis in affected knee

Exclusion Criteria:

* intraarticular corticosteroids in affected knee within past three months
* primary inflammatory connective tissue disease (ie rheumatoid arthritis)
* currently taking oral corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kalunian, MD, Principal Investigator — University of California, San Diego; Anna Quan, MD, Study Chair — San Diego VA Hospital; Michal Kalli Hose, MD, Study Director — San Diego VA Hospital; Jeannie Chao, MD, Study Director — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego Medical Center, La Jolla, California
  - San Diego VA Hospital, La Jolla, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in rheumatology clinics at UCSD and the VA musculoskeletal clinic.
Pre-assignment Details: Patients taking oral corticosteroids, who had a primary inflammatory connective tissue disease, or who received IA corticosteroids in the affected knee within three months of study entry were excluded from the study.
Groups:
- Placebo: Intraarticular injection of 0.9% saline
Period: Overall Study
Arm/Group | Corticosteroid Injection | Placebo
Started | 40 | 39
Completed | 36 | 35
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroid Injection | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 16 | 16 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (12) | 63 (12) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 39 | 37 | 76
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change in Western Ontario and McMasters Universities Arthritis Index (WOMAC) Pain Subscale
Description: WOMAC pain subscale range 0-20 (0=best, 20=worst)
Time Frame: baseline to 4 weeks
Population: This population was defined as patients who completed the 4 week follow up assessment as per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Corticosteroid Injection | Placebo
Number analyzed (Participants) | 33 | 34
units on a scale | -2.1 (2.6) | -0.1 (1.9)

2. Other Pre Specified Outcome: Change in WOMAC Pain Subscale
Description: WOMAC pain subscale range 0-20 (0=best, 20=worst)
Time Frame: baseline to 12 weeks
Population: These patients were categorized as inflammatory or noninflammatory based on the baseline ultrasound characteristics. All patients were in the treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Inflammatory Patients Who Received Corticosteroid Injections: Patients with inflammatory characteristics on ultrsaound who were treated with corticosteroid knee injections
- Noninflammatory Patients Who Received Corticosteroid Injection: Patients with noninflammatory characteristics on ultrasound who received saline placebo knee injections
Arm/Group | Inflammatory Patients Who Received Corticosteroid Injections | Noninflammatory Patients Who Received Corticosteroid Injection
Number analyzed (Participants) | 16 | 14
units on a scale | -0.1 (3.2) | -2.0 (1.8)

ADVERSE EVENTS:
Arm/Group | Corticosteroid Injection | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No